CLINICAL TRIAL: NCT02990819
Title: Phase II Study for Patients With Primary Immunodeficiencies Using and Cd19+ Depleted Unrelated Donor or Partially Matched Related Donor Peripheral Stem Cells
Brief Title: Alpha/Beta T and CD19+ Depleted Peripheral Stem Cells for Patients With Primary Immunodeficiencies
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Timothy Olson, Medical Director, Hematopoietic Stem Cell Transplantation (HSCT) Program, Children's Hospital of Philadelphia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-011733; 15BT022 (Other: CHOP)
Record Dates: First submitted 2016-12-05; First posted 2016-12-13 (Estimated); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Immunodeficiencies; Immune Dysregulation Syndromes
Keywords: Immunodeficiencies; Immune dysregulation syndromes
MeSH Terms: conditions — Immunologic Deficiency Syndromes

STUDY DESIGN:
Intervention Model Description: T-depleted stem cell infusion
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Reduced intensity regimen (Other): Conditioning regimen is dependent on patient diagnosis and age. Reduced intensity conditioning with chemotherapy followed by stem cell transplant using the CliniMACs device to deplete alpha/beta T and CD19+ peripheral stem cells. Standard of care reduced intensity conditioning will include Busulfan, Fludarabine, Thiotepa followed by stem cell infusion.
  Interventions: Device: Apha/beta T and CD19+ cell depletion using CliniMACS device
- Myeloablative regimen (Other): Conditioning regimen is dependent on patient diagnosis and age. Patients with chronic granulomatous disease or Wiskott-Aldrich syndrome will receive cyclophosphamide in lieu of thiotepa to ensure engraftment.
  Myeloablative regimen with chemotherapy followed by stem cell transplant using the CliniMACs device to deplete alpha/beta T and CD19+ peripheral stem cells. Standard of care myeloablative regimen will include Busulfan, Fludarabine, Thiotepa, or Cyclophosphamide followed by stem cell infusion.
  Interventions: Device: Apha/beta T and CD19+ cell depletion using CliniMACS device
- Immunotherapy (Other): Conditioning regimen is dependent on patient diagnosis and age. Severe combined immunodeficiency (SCID) patients will be conditioned with immunotherapy only followed by stem cell transplant using the CliniMACs device to deplete alpha/beta T and CD19+ peripheral stem cells. Immunotherapy regimen will include anti-thymocyte globulin followed by stem cell infusion.
  Interventions: Device: Apha/beta T and CD19+ cell depletion using CliniMACS device

INTERVENTIONS:
Device: Apha/beta T and CD19+ cell depletion using CliniMACS device — Stem cells will be processed using the CliniMACS device for alpha/beta and CD19+ T cell depletion. Processing of cells using the CliniMACS will occur in accordance with the Investigator Brochure and Technical Manual following the laboratory standard operating procedures (SOPs) and using aseptic technique.

SUMMARY:
This is a Phase II trial to determine the ability of a reduced intensity conditioning regimen to allow successful engraftment with alpha/beta T and CD19+ depleted peripheral stem cell grafts from unrelated or partially matched related donors. There are two conditioning regimens depending upon patient diagnosis and age.

DETAILED DESCRIPTION:
This is a Phase II trial to determine the ability of a reduced intensity conditioning regimen to allow successful engraftment with alpha/beta T and CD19+ depleted peripheral stem cell grafts from unrelated or partially matched related donors. There are two conditioning regimens depending upon patient diagnosis and age.

The study will include patients 0-25 years with PID, including immune dysregulation syndromes for which hematopoietic stem cell transplant is indicated.

Treatment: Either conditioning regimen (listed below) followed by alpha/beta T and CD19+ depleted donor peripheral stem cells

1. Reduced intensity conditioning with busulfan x 8 doses, fludarabine 40 mg/m2 x 4, thiotepa 5 mg/kg x 2, anti-thymocyte globulin (ATG) 3 mg/kg x 3.

   OR
2. Myeloablative regimen with busulfan x 16 doses or Daily for four days, fludarabine 30 mg/m2 x 5, thiotepa 5 mg/kg x 2, ATG 3 mg/kg x 2.

   OR
3. Immunotherapy regimen on days -9, 8, 7 with anti-thymocyte globulin 3 mg/kg/day (for severe combined immunodeficiency patients only).
4. Infusion of alpha/beta T and CD19+ depleted donor peripheral stem cells.
5. Follow up, including evaluation of chimerism and immune reconstitution.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 0-25 years at time of enrollment
2. Diseases:

   * Immunodeficiencies for which allogeneic hematopoietic stem cell transplant is indicated, including severe combined immunodeficiencies, immunodeficiency polyendocrinopathy X-linked syndrome (IPEX), X-linked lymphoproliferative disease, chronic granulomatous disease, Wiskott-Aldrich syndrome (WAS), hyperIgM, and other life-threatening immunodeficiencies.
   * Immune dysregulation syndromes, including refractory or recurrent hemophagocytic lymphohistiocytosis, hemophagocytic lymphohistiocytosis (HLH) with genetic mutations, refractory multisystemic Langerhans cell histiocytosis, other macrophage activating syndrome (MAS) refractory to standard therapy.
3. Clinical status

   * Lansky or Karnofsky performance >=60
   * Organ Function:

     1. Serum creatinine <1.5 x upper limit of normal for age Hepatic: ALT <=250; AST <=350
     2. Cardiac shortening fraction >=27%
     3. Bilirubin <2.5x normal (unless elevation due to Gilberts disease).
     4. No active untreated infection
4. Signed informed consent
5. No HLA matched related donor available.
6. Females of childbearing potential must have negative pregnancy test.

Exclusion Criteria:

* Uncontrolled bacterial, viral or fungal infections
* HLA matched related or unrelated donor able to donate mobilized peripheral stem cells.
* Pregnant Females
* Matched related donor available for bone marrow donation

Donors Selection Criteria:

* Donor selection will comply with 21 CFR 1271
* Unrelated donor matched or up to one antigen mismatch as per National Marrow Donor Program (NMDP).
* Haploidentical parent or sibling able to undergo mobilization for peripheral stem cell collection. Maternal donor preferred over paternal donor if both equally haploidentical.
* Children's Hospital of Philadelphia (CHOP) Blood and Marrow Transplant (BMT) procedures apply for determining donor eligibility, including donor screening and testing for relevant communicable disease agents and diseases.
* Unrelated donor identified through the National Marrow Donor Program (NMDP) and fulfills the NMDP criteria for donation. Unrelated donor willing and able to undergo mobilization of peripheral stem cells and apheresis

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-12; Primary Completion 2026-11 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Event free survival | One year
  Event free survival in greater than 20 percent donor cells at one year for patients with primary immunodeficiencies (PID) who receive unrelated or partially matched related donor peripheral stem cell grafts which have been alpha/beta T depleted and CD19 depleted
Stable engraftment | One year
  Stable engraftment in greater than 20 percent donor cells at one year for patients with primary immunodeficiencies (PID) who receive unrelated or partially matched related donor peripheral stem cell grafts which have been alpha/beta T depleted and CD19 depleted

SECONDARY OUTCOMES:
Severity of graft vs. host disease (GVHD) | One and two years
  Severity of acute and chronic graft vs host disease (GVHD), incidence of mixed chimerism, primary and secondary graft rejection, and immune reconstitution at one and two years
Incidence of graft vs. host disease (GVHD) | One and two years
  Evaluation of incidence of chronic graft vs host disease (GVHD), incidence of mixed chimerism, primary and secondary graft rejection, and immune reconstitution at one and two years

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Olson, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No